CLINICAL TRIAL: NCT02650726
Title: Effect of Purification Anthocyanins on HDL and Endothelial Function in Subjects With Type 2 Diabetes Mellitus: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Purified Anthocyanins Supplementation and High-Density Lipoprotein (HDL) Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Di Li, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZXYZM-4
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus，Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): The participants in this group are instructed to consume placebo capsules every day during the trial period.
  Interventions: Other: Placebo
- treatment group (Experimental): The participants in this group are instructed to consume anthocyanin capsules every day during the trial period.
  Interventions: Dietary Supplement: Anthocyanin

INTERVENTIONS:
Dietary Supplement: Anthocyanin — anthocyanin 320 mg daily for 24 weeks
  Other Names: MEDOX (natural purified anthocyanin)
  Arms: treatment group
Other: Placebo — placebo 320mg daily for 24 weeks
  Arms: control group

SUMMARY:
HDL function is impaired in patients with type 2 diabetes mellitus. Anthocyanin, a water-soluble compounds,is beneficial for vascular function by increasing nitric oxide (NO) bioavailability and decreasing oxidative stress. This study was designed to evaluate whether anthocyanin supplementation might improve cardiovascular function in diabetic patients.

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blind label, interventional study on patients with T2DM. The eligible participants are randomly assigned to control and anthocyanins group. During the 24 weeks trial period, the participants are instructed to consume two anthocyanin capsules or placebo capsules twice daily (30 minutes after breakfast and supper).

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with type 2 diabetes mellitus according to the Chinese type 2 diabetes prevention guide 2010, diagnostic criteria are as follows: (1) Diabetes symptoms（polydipsia、polyphagia, polyuria, weight loss、skin itching、blurred vision and other acute metabolic network disorder that caused by high blood sugar）combined with random blood sugar ≥11.1 OR, (2) fasting plasma glucose (FPG) ≥7.0 OR, (3) 2 h blood sugar after oral glucose tolerance test (OGTT) ≥11.1
* Subject is between 40 and 60 years of age, inclusive
* Subject's BMI is >18.5 kg/m2 and <35 kg/m2.

Exclusion Criteria:

* Subject that is diagnosed as type 1 diabetes, gestational diabetes and other kinds of diabetes expect type 2
* Subject that is pregnant
* Subject that has coronary artery disease, mental disorder, cancer, cirrhosis, renal disease and hepatic disease
* Subject that has had operation less than six months prior to screening visit
* Subject that uses multivitamin supplement or other polyphenol supplement

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
HDL-associated PON1 activity | 24 weeks
  PON1 activity is assayed in HDL isolated from plasma of subjects from the placebo and anthocyanin groups by using UV spectrophotometry in a 96-well plate format using phenyl acetate or paraoxon as substrates.
The anti-oxidative ability of HDL | 24 weeks
  The anti-oxidative ability is assayed in HDL isolated from plasma of subjects from the placebo and anthocyanin groups by using fluorescence measurement in a 96-well plate format using dihydrorhodamine(DHR) as substrates.
anti-inflammatory ability of HDL | 24 weeks
  The ability of anti-inflammatory ability of HDL is showed as HDL inflammatory index (HII).HII means the ability of apolipoprotein (apo)B-depleted serum to inhibit or enhance the oxidation of LDL in the presence of a fluorescent organic phospholipid 2',7'-dichlorodihydrofluorescein diacetate (DCF) fluoresces substrate.

SECONDARY OUTCOMES:
endothelium-dependent flow-mediated dilatation (FMD) | 24 weeks
  Endothelial function as determined by the flow-mediated dilatation (FMD) and endothelium-independent glyceryltrinitrate-induced dilation (GTND) were measured noninvasively in the right brachial artery by use of a high-resolution ultrasound scanning echo-tracking angiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Di Li, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guangdong Provincial Key Laboratory of Food, Nutrition and Health, Department of Nutrition, School of Public Health, Sun Yat-Sen University (Northern Campus), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
It depends on the Sponsor Investigator